CLINICAL TRIAL: NCT06191874
Title: Evaluation of Advanced Imaging and Visualization to Clinical Deep Brain Stimulation
Brief Title: Evaluation of Advanced Imaging and Visualization for Clinical Deep Brain Stimulation
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00113490; R37NS116079 (NIH)
Record Dates: First submitted 2023-12-06; First posted 2024-01-05 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-02

CONDITIONS: Deep Brain Stimulation
Keywords: DBS; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery planning by SOC methods, then by HoloDBS: Standard-of-care (SOC) surgery plan is built before the HoloDBS hypothetical surgery plan
  Interventions: Other: Standard-of-care (SOC) surgery plan; Other: HoloDBS hypothetical surgery plan
- Surgery planning by HoloDBS, then by SOC methods: HoloDBS hypothetical surgery plan is built before the standard-of-care (SOC) surgery plan
  Interventions: Other: Standard-of-care (SOC) surgery plan; Other: HoloDBS hypothetical surgery plan

INTERVENTIONS:
Other: Standard-of-care (SOC) surgery plan — Use of SOC clinical planning tools to prepare for DBS (deep brain stimulation) surgery
Other: HoloDBS hypothetical surgery plan — Use of next generation visualization tools and surgical targeting models to hypothetically prepare for DBS (deep brain stimulation) surgery

SUMMARY:
The objective of this project is to evaluate next generation visualization tools and surgical targeting models for clinical deep brain stimulation (DBS).

This study will evaluate the performance of HoloDBS software in comparison to the current standard (SOC) clinical planning tools to prepare for DBS surgery. The investigators hypothesize that HoloDBS will provide more detailed and anatomically useful information to the neurosurgeon and neurologist than the current clinical standard.

The study team reviews electronic medical records (EMR) from patients who are undergoing DBS surgery. There are no study visits involved in this study as only data from standard clinical care will be used. All study activities are executed by the study team and there are no interventions.

ELIGIBILITY:
Electronic medical records (EMR) from all patients undergoing preoperative DBS evaluation will be reviewed and their data will be used for this study's purposes if they fit the inclusion and exclusion criteria.

Inclusion criteria:

* age 18 years and over
* meeting qualification for deep brain stimulation for Parkinson's disease with one or more of medication refractory tremor, motor fluctuations despite medication optimization, or levodopa responsiveness but limited by medication induced adverse effects (nausea, dystonia, dyskinesia for example).

Exclusion criteria:

* consideration of alternate diagnosis to Parkinson disease
* high risk medical comorbidities which would make the patient not a candidate for surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease scheduled for Deep Brain Stimulation Surgery
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Difference between the actual post-operative location of the DBS electrode and the planned location. | 1 month after surgery
  Comparison of the post-operative position of the DBS electrode to the location that was defined in the standard-of-care plan and the HoloDBS plan.

SECONDARY OUTCOMES:
Number of physicians who reply 'yes' to the question, 'Was the additional data available in the HoloDBS application valuable in defining your theoretical optimal electrode position?' | 6 months and 1 year after study starts
  Open ended discussion with neurosurgery-neurology team

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No